CLINICAL TRIAL: NCT02454686
Title: Role of Fibroscan in Predicting Complications After Hepatectomy
Brief Title: Fibroscan Predicts Complications After Hepatectomy
Acronym: Fibroscan
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Prof. Guido Torzilli, Professor of Surgery, University of Milan
Other Study IDs: Fibroscan
Record Dates: First submitted 2015-05-19; First posted 2015-05-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Liver Neoplasms
Keywords: Complications after hepatectomy
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Most of the postoperative complications that may occur after hepatectomy are related to the underlying liver background, and the common preoperative tests do not completely predict such complications. Transient elastography by Fibroscan is used to calculate the stiffness and the steatosis of the liver, and it may be also used to predict postoperative complications after hepatectomy

DETAILED DESCRIPTION:
A prospective cohort study on consecutive patients scheduled for hepatectomy was planned. Fibroscan was performed during the preoperative workup. Accuracy of the liver stiffness and steatosis measured by Fibroscan in predicting the presence of cirrhosis, of steatosis, and the development of postoperative complications was assessed by ROC curve, and multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary and secondary tumors scheduled for hepatectomy at our Unit
* Written consent to get the Fibroscan during the preoperative workup

Exclusion Criteria:

* Refute to get the Fibroscan
* Loss of data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective cohort of patients scheduled for hepatectomy.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2012-02; Primary Completion 2014-10 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Accuracy of Fibroscan in predicting complication after hepatectomy | 90 days
  Calculation of the accuracy of the liver stiffness and steatosis measured with the Fibroscan in predicting complications after hepatectomy. The values of the stiffness and steatosis will be correlated with the number of complications

CONTACTS AND LOCATIONS:
Overall Officials: Guido Torzilli, MD, PhD, Study Director — Humanitas Research Hospital IRCCS, Rozzano-Milan

REFERENCES:
- [Derived] Donadon M, Fontana A, Palmisano A, Vigano L, Procopio F, Cimino M, Del Fabbro D, Torzilli G. Individualized risk estimation for postoperative morbidity after hepatectomy: the Humanitas score. HPB (Oxford). 2017 Oct;19(10):910-918. doi: 10.1016/j.hpb.2017.06.009. Epub 2017 Jul 22. PMID 28743491